CLINICAL TRIAL: NCT06383507
Title: A Phase I Clinical Study to Assess the Safety and Efficacy of CD70-targeted CAR-T in the Treatment of CD70-positive Refractory or Relapsed Solid Tumors
Brief Title: A Clinical Study of Anti-CD70 UCAR-T in Relapsed or Refractory Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT101
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Tumor; Advanced Solid Tumor; Renal Cell Carcinoma; Ovarian Cancer; Cervix Cancer; Head and Neck Squamous Cell Carcinoma; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Renal Cell; Ovarian Neoplasms; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD70 UCAR-T Cell Injection (Experimental): In the discovery phase, accelerated titration combined with the "3+3" dose escalation principle was adopted, starting from the initial dose of 3×106/kg. If a grade ≥3 AE occurs during DLT observation, the accelerated titration mode will switch to "3+3" dose escalation, at least 12 eligible patients will be enrolled and receive 4 doses of CD70 UCAR-T cell therapy (3 × 10^6 cells/kg, 6 × 10^6 cells/kg, 8× 10^6 cells/kg, 1 × 10^7 cells/kg).
  In the dose expansion phase, each group will choose one or two dose groups to verify the safety and efficacy, and plan to recruit about 6 subjects in each dose group.
  Interventions: Drug: CHT101

INTERVENTIONS:
Drug: CHT101 — After lymphodepletion with Fludarabine and Cyclophosphamide, CD70 UCAR T cells were transfused intravenously.

SUMMARY:
This is a single-center, single-arm ，open-label ，dose escalation and dose extension study. In this study we plan to evaluate the safety and efficacy of CD70-targeting UCAR-T cells in the treatment of CD70-positive refractory or relapsed solid tumors, and obtain recommended doses and infusion patterns.

DETAILED DESCRIPTION:
In the discovery phase, accelerated titration combined with the "3+3" dose escalation principle was adopted, starting from the initial dose of 3×106/kg. If a grade ≥3 AE occurs during DLT observation, the accelerated titration mode will switch to "3+3" dose escalation, at least 12 eligible patients will be enrolled and receive 4 doses of CD70 UCAR-T cell therapy (3 × 10^6 cells/kg, 6 × 10^6 cells/kg, 8× 10^6 cells/kg, 1 × 10^7 cells/kg).

In the dose expansion phase, each group will choose one or two dose groups to verify the safety and efficacy, and plan to recruit about 6 subjects in each dose group.

During the clinical study, after the completion of each dose group, the Safety Monitoring Committee (SMC) will determine whether it is possible to continue to increase to the next higher dose group, or add more subjects to the current dose group, or reduce to a lower dose group to continue to explore, or climb to a higher dose after reaching the highest dose (1 × 10^7 cells/kg).

Conditions Relapsed Tumor, Refractory Solid Tumor, Renal Cell Carcinoma, Head and Neck Squamous Cell Carcinoma, Nasopharyngeal carcinoma, Ovarian Cancer, Cervix Cancer etal

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign a written informed consent documen；
2. Age ≥18 years old, male or female；
3. Histopathological confirmed advanced or metastatic solid tumors failed to at least second-line treatment or initially diagnosed advanced/metastatic solid tumors that have no NCCN guideline recommended standard first-line therapy；
4. Histopathology or cytology (paraffin section or fresh biopsy tumor tissue specimen) diagnosed as advanced/metastatic solid tumor (positive tumor CD70 expression (tumor CD70 positive (IHC 2+) confirmed by histology or pathology));
5. At least one measurable lesion at baseline per RECIST version 1.1；
6. The expected survival time is more than 12 weeks;
7. ECOG 0-1 points;
8. The function of important organs is basically normal:Hematopoietic function:

   * Hematopoietic function: neutrophils ≥ 1.5×109/L, platelets ≥ 90×109/L, hemoglobin ≥ 90g/dL;
   * Renal function: serum creatinine≤1.5×ULN;
   * WBC≥3.0×109/L,
   * Liver function: Total bilirubin ≤ 1.5×ULN(Except Gilbert syndrome), extrahepatic metastasis：ALT and AST ≤ 3.0×ULN (Nonhepatic metastasis：it can be relaxed to ≤ 5.0×ULN);
   * coagulation function：INR≤1.5×ULN，APTT≤1.5×ULN
9. Subjects agree to use reliable and effective contraceptive methods for contraception within 6 months after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception);

Exclusion Criteria:

1. Received anti-CD70 drug treatment before screening;
2. Received anti-tumor therapy such as chemotherapy and targeted therapy within 2 weeks or at least 5 half-lives (whichever is longer) before Received;
3. Received systemic corticosteroid therapy at doses greater than 10 mg/day prednisone (or equivalent doses of other corticosteroids) within 2 weeks prior to Received；
4. Pregnant, lactating, or breastfeeding females;
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Virus (HCV) RNA titer test is greater than the normal range; human immunodeficiency virus (HIV) antibody positive; syphilis test positive; cytomegalovirus (CMV) DNA test positive;
6. Have any of the following heart conditions:

   New York Heart Association (NYHA) stage III or IV congestive heart failure; Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment; Clinically significant ventricular arrhythmia, echocardiography showed cardiac ejection fraction<50%,
7. Active/symptomatic central nervous system metastases or meningeal metastases at the time of screening; subjects with brain metastases who have been treated must be confirmed to have no imaging evidence of progression ≥ 4 weeks after the end of treatment before they can be enrolled;
8. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation;
9. Vaccination within 14 days of study enrollment;
10. Received live attenuated vaccine within 4 weeks before screening;
11. Malignant tumors other than the target tumor within 3 years prior to screening, except for the following: malignant tumors that have received radical treatment and no known active disease within ≥ 3 years prior to enrollment;
12. Other investigators deem it inappropriate to participate in the study.
13. Serious or uncontrollable systemic disease or any unstable systemic disease, including but not limited to uncontrolled hypertension, uncontrolled hyperglycemia, liver and kidney insufficiency or metabolic disease, central nervous system disease, etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2027-04-21 (Estimated); Study Completion 2029-04-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CD70 UCAR-T cells infusion (Safety and Tolerability) | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Disease control rate (DCR) | 42 days
  The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Objective response rate (ORR) | 42 days
  The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.

IPD SHARING:
Plan to Share IPD: No